CLINICAL TRIAL: NCT02261974
Title: VIveve Treatment of the Vaginal Introitus to EValuate Effectiveness
Acronym: VIVEVE I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viveve Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: (OUS) V-013
Record Dates: First submitted 2014-09-29; First posted 2014-10-10 (Estimated); Results first posted 2017-12-27 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Vaginal Laxity Following Childbirth; Sexual Function Following Childbirth
Keywords: Vaginal laxity; Sexual Function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Viveve Treatment (Active Comparator): Intervention in the active arm will be with the Viveve System using 90 Joules/cm2 active treatment with radiofrequency energy in the vaginal introitus
  Interventions: Device: Active Treatment Viveve
- Sham Viveve Treatment (Placebo Comparator): Intervention in the sham arm will be with the Viveve System using ≤1 Joule/cm2 sham treatment with radiofrequency energy in the vaginal introitus
  Interventions: Device: Sham Treatment Viveve

INTERVENTIONS:
Device: Active Treatment Viveve — Subject will receive 90 Joules/cm2 radiofrequency energy to the vaginal introitus
  Arms: Active Viveve Treatment
Device: Sham Treatment Viveve — Subject will receive ≤ one (1) Joule of radiofrequency energy to the vaginal introitus
  Arms: Sham Viveve Treatment

SUMMARY:
Outside United States (OUS) Post-Market Parallel Group Exploratory Study Design

The objective of this study is to determine the safety and effectiveness of the Viveve System to treat the vaginal introitus in women following vaginal birth(s) and in so doing improving vaginal laxity.

DETAILED DESCRIPTION:
A prospective, longitudinal, randomized, single-blind, sham controlled clinical study is planned. This study is designed to demonstrate that the active treatment (i.e., Viveve Procedure) is superior to the sham treatment for the primary effectiveness and safety endpoints.

Approximately 113 evaluable subjects will be randomized in a 2:1 ratio to either the active treatment group or sham group. The active treatment group will receive a treatment dose of 90 J/cm2 and the sham group will receive a sub-treatment dose of ≤1 J/cm2.

Subjects will be followed up at 72 hrs, 10 days, and one, two, three, and six months post treatment.

Final data will be reported at 6 months for active and sham treatments.

ELIGIBILITY:
Key Inclusion Criteria:

1. Able to understand and voluntarily sign the informed consent form
2. Pre-menopausal and ≥ 18 years of age
3. At least one full term vaginal delivery (> 37 completed weeks gestation) at least 12 months prior to enrollment date
4. Experiences vaginal looseness (laxity) during vaginal intercourse
5. Subject must have a screening blood count and metabolic panel including FSH level of <35 mIU/mL (35 IU/L).
6. Subject must have a normal pelvic exam at baseline and negative chlamydia and gonorrhea cultures during the screening period.
7. Subject had a normal PAP within last three years, cytology, no HPV and within last five years, cytology and no HPV.
8. Subject must be willing to engage in vaginal intercourse at least once per month.
9. Subject must be in a monogamous, heterosexual relationship for at least six months prior to screening visit with a partner who is sexually functional and available at least 50% of the time.
10. Subject is surgically sterilized, or is willing to use an acceptable method of birth control that was begun at least 3 month prior to screening and to be continued or throughout the duration of the study [i.e., barrier method (e.g., diaphragm), hormonal therapy (subcutaneous, injectable, or oral contraceptive) intrauterine device], or partner is surgically sterilized

Key Exclusion Criteria:

1. Pregnant or planning to become pregnant within the next 12 months or has had a delivery within the last 12 months.
2. Currently breastfeeding or discontinued breast feeding fewer than 6 months prior to enrollment
3. History of a genital fistula, a thin recto-vaginal septum as determined by the investigator, or history of a fourth degree laceration during screening physical exam
4. Clinically significant pelvic organ prolapse
5. Currently meets the criteria for a female sexual disorder, including DSM V, FSAD, FOD, Genitopelvic Pain, Sexual Aversion, Dyspareunia, or Vaginismus, and has not been treated for this condition within the past 12 months
6. Beck Depression Inventory score > 14
7. DSM-5 psychiatric diagnosis exhibiting clinically significant symptoms
8. Taking SSNRI or SSRI drugs
9. Not willing to abstain from vaginal intercourse or use of tampons until 10-day follow-up visit completed
10. Evidence of active sexually transmitted disease upon vaginal exam that precludes treatment
11. History of genital herpes
12. Clinically significant abnormalities in clinical chemistry or hematology at the time of screening
13. Currently taking prescribed medications, OTC products or supplements that may impact or enhance sexual function (e.g., antihypertensive, psychotropic, chemotherapeutic agent, PD5 Inhibitors) as assessed by the investigator
14. Currently undergoing chemotherapy, radiation therapy, or pelvic floor physical therapy
15. Has an implantable pacemaker, an automatic implantable cardioverter/defibrillator (AICD), or any other implantable electrical device, as these devices may be adversely affected by radiofrequency fields or current
16. Has undergone the Viveve Procedure previously
17. Has medical condition that in investigator's opinion may interfere with wound healing response
18. Has an acute or a chronic vaginal or vulvar disorder (e.g., vaginal atrophy, pain including vulvodynia, vulvar vestibulitis dysethetic vulvodynia or vulvar dystrophy, current/chronic papulosquamous vulvar dermatoses (e.g., psoriasis lichen planus, tinea cruris, lichen sclerosis, seborrhea dermatitis, contact or irritant dermatitis, lichen simplex, eczema) or bullous dermatoses or systemic diseases with potential involvement of vulva)
19. Has Irritable Bowel Syndrome or Crohn's Disease
20. Has dyspareunia defined as recurrent or persistent painful intercourse that affects sexual activity
21. Has been in another clinical study within four weeks of screening, or is not willing to abstain from enrolling in other clinical studies for duration of trial

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Wilkerson, PhD, Study Director — Viveve Inc.
Locations (9):
- Canada (4):
  - Allan Centre, Calgary, Alberta
  - Complexe Medical St-Laurent, Montreal, Quebec
  - Les Cours Medical Centre, Montreal, Quebec
  - Exogenia Institute of Anti-Aging and Regenerative Medicine, Sherbrooke
- Research Center of Reproductive Medicine. - IRCCS Policlinico San Matteo Hospital, Pavia, Italy
- Japan (2):
  - Yokohama Motomachi Jyosei Iryou Clinic Luna, Kanagawa
  - Naoe Beauty Clinic, Tokyo
- Spain (2):
  - Instituto Palacios, Salud de la Mujer, Madrid
  - Unidad de Gestión Clínica de Obstetricia y Ginecología. Hospital Universitario Araba, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Viveve Treatment | Sham Viveve Treatment
Started | 123 | 63
Treated | 117 | 57
Completed | 108 | 56
Not Completed | 15 | 7
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Missed treatment cut-off date | 6 | 3
Not completed — Received partial treatment; FU to 1 mo | 3 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Viveve Treatment | Sham Viveve Treatment | Total
Number analyzed (Participants) | 123 | 63 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (6.0) | 41.1 (5.6) | 40.8 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 63 | 186
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (4.6) | 24.4 (5.4) | 24.5 (4.8)
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 7 | 2 | 9
  Ear, nose, or throat condition | 6 | 7 | 13
  Dermatologic condition | 9 | 4 | 13
  Pulmonary condition | 2 | 4 | 6
  Hepatic or biliary condition | 3 | 4 | 7
  Endocrine condition | 12 | 5 | 17
  Neurologic condition | 10 | 3 | 13
  Psychiatric condition | 3 | 3 | 6
  Hematologic condition | 8 | 5 | 13
  Allergies | 20 | 13 | 33
  Gynecologic condition | 19 | 7 | 26
  Prior Surgeries | 82 | 41 | 123
  Prior STD | 7 | 2 | 9
Gravidity Per Subject [Mean (Standard Deviation); unit: Pregnancies] — Average number of reported pregnancies per subject
  Pregnancies | 2.7 (1.4) | 2.7 (1.3) | 2.7 (1.4)
Time Since Last Delivery [Mean (Standard Deviation); unit: years] | 8.0 (6.3) | 8 (5.5) | 8 (6)
Median Birth weight [Mean (Standard Deviation); unit: kg] — Maternal History: Average of median birth weights.
  kg | 3.3 (.7) | 3.4 (.5) | 3.3 (.6)
Number of Vaginal Deliveries per Subject [Mean (Standard Deviation); unit: Number of Reported Vaginal Deliveries] | 2.1 (1) | 2 (.9) | 2.1 (.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Female Sexual Function Index (FSFI) Total Score
Description: The mean change from baseline in FSFI total score in the active arm compared to the sham arm. The FSFI is a 19-item validated measure of female sexual function. It consists of 6 domains: Desire, Arousal, Lubrication, Orgasm, Satisfaction, and Pain. Each item's score can range from 0-5 (or 1-5 in several instances). For individual domain scores, the scores of the individual items that comprise the domain are summed, and the sum is multiplied by the domain factor (factors are permanent and do not change). The 6 domain scores are then summed to obtain the FSFI total score. The total score ranges from 2-36. A higher score indicates a greater level of sexual function, while a lower score correlates to a greater level of sexual dysfunction. Within individual domains, a domain score of 0 indicates that the subject reported having no sexual activity during the past month. The baseline score is the FSFI total score from the screening visit.
Time Frame: 6 months
Population: This population consists of all randomized subjects who completed the six month assessment.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Active Viveve Treatment | Sham Viveve Treatment
Number analyzed (Participants) | 108 | 55
Units on a Scale | 4.16 (0.48) | 2.36 (0.67)

2. Primary Outcome: Reporting Adverse Events (AEs)
Description: Proportion of subjects in the active arm relative to those in the sham arm experiencing a treatment-related AE by six months post-intervention.
Time Frame: 6 months
Population: Table includes treatment-emergent adverse events (AEs), defined as AEs that began or worsened in severity after treatment.
  This population consists of all subjects who were randomized and who received a complete or partial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Viveve Treatment | Sham Viveve Treatment
Number analyzed (Participants) | 117 | 57
Participants | 13 | 7

3. Secondary Outcome: Mean Change From Baseline in Vaginal Introitus Laxity Inventory (VALI) Total Score
Description: Vaginal Introitus Laxity Inventory (VALI) is a 12-item patient reported outcome measure designed to describe and quantify the nature of a female respondent's concern with the perception of laxity ("looseness") and its impact on the qualities of satisfaction and enjoyment of her sexual functioning. Items of the VALI address the impact of laxity on the major aspects of the female sexual response cycle (i.e., sexual desire, arousal and orgasm), and quantify the patient's experience of sexual pleasure, sensitivity and satisfaction. The VALI items also address the potential impact of vaginal introitus laxity on sexual confidence and the patient's partner. All 12 items are measured on 5-point Likert scales (0= Very Poor, 1=Poor, 2=Moderate, 3=Good, 4=Very Good) and scores are summed to achieve a VALI Total score, range 0-48. A higher score corresponds to positive sexual satisfactions and functioning.
Time Frame: 6 months
Population: This population consists of all randomized subjects with a 6 month assessment.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Active Viveve Treatment | Sham Viveve Treatment
Number analyzed (Participants) | 107 | 56
Units on a Scale | 7.28 (0.64) | 6.32 (0.89)

4. Secondary Outcome: Mean Change From Baseline in the VSQ Vaginal Laxity Question (VLQ)
Description: Mean change in VSQ Vaginal Laxity Question (VLQ) score from baseline to 6 months post-intervention. The VLQ is one question. The global assessment of vaginal laxity is scored on a seven-point Likert type scale where the response to the question ranges from 1-7 where 1 = "Very Loose" and 7 = "Very Tight". The Likert-scale is one of the most widely used bipolar scaling method instruments in survey research. The VSQ VLQs levels of vaginal laxity uses a balanced keying (an equal number of positive and negative statements) to obviate the problem of acquisition bias. Baseline VLQ is the score indicated that the screening visit.
Time Frame: 6 months
Population: This population consists of all randomized subjects who completed a 6 month assessment.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Active Viveve Treatment | Sham Viveve Treatment
Number analyzed (Participants) | 108 | 56
Units on a Scale | 1.81 (0.15) | 1.07 (.21)

5. Secondary Outcome: Mean Change From Baseline in Female Sexual Distress Scale - Revised (FSDS-R)
Description: The mean change in total FSDS-R score from baseline to six months post-intervention in the active arm compared to the sham arm. The FSDS-R is a 12-item patient-reported questionnaire and a validated scale used to measure sexually-related personal distress in women. Women rate 13 questions as Never (0), Rarely (1), Occasionally (2), Frequently (3), and Always (4), for a total score range of 0-52 (the individual question scores are summed to give the total score). A higher frequency of occurrences (which correlates to a total higher score) indicates a greater distress or a "worse outcome". The numbers below represent the changes from baseline in mean FSDS-R total score. The baseline value is the FSDS-R total score at screening.
Time Frame: 6 months
Population: This population consists of all randomized subjects who completed a 6 month assessment.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Active Viveve Treatment | Sham Viveve Treatment
Number analyzed (Participants) | 107 | 56
Units on a Scale | -6.55 (0.74) | -4.13 (1.02)

ADVERSE EVENTS:
Time Frame: 6 months post-treatment
Description: The definitions of adverse event (AE) and serious adverse event (SAE) used in this study were consistent with the clinicaltrials.gov definitions. Severity was graded using Common Terminology Criteria for Adverse Events (CTCAE), Version 4.3, which stratifies severity across five (5) levels rather than the three (3) used in the clinicaltrials.gov definitions.
Arm/Group | Active Viveve Treatment | Sham Viveve Treatment
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/117 | 1/57
Other Adverse Events (participants affected / at risk) | 38/117 | 20/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Viveve Treatment (N=117) | Sham Viveve Treatment (N=57)
Kidney Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Viveve Treatment (N=117) | Sham Viveve Treatment (N=57)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 2 (2) | 1 (1)
Inflammation (General disorders) | 1 (1) | 1 (1)
Polyp (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bacterial Vaginosis (Infections and infestations) | 2 (2) | 1 (1)
Candida Infection (Infections and infestations) | 1 (1) | 2 (2)
Chlamydial Infection (Infections and infestations) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Genital Herpes Simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Mycoplasma Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 4 (5) | 3 (3)
Vaginal Infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0)
Sports Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Helicobacter Test Positive (Investigations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Facial Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Coital Bleeding (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypomenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Inadequate Lubrication (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Premenstrual Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pruritus Genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Uterine Spasm (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal Discharge (Reproductive system and breast disorders) | 5 (6) | 2 (2)
Vulval Disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal Burning Sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulvovaginal Dryness (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulvovaginal Erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal Swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No